CLINICAL TRIAL: NCT06380478
Title: Safety and Efficacy of the Bi-Aspheric Monofocal Intraocular Lens
Brief Title: Safety and Efficacy of the Bi-Aspheric Monofocal IOL
Status: Recruiting | Type: Observational
Sponsor: ICARES Medicus, Inc. (Industry)
Collaborators: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPRO-000012
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: Cataract; Monofocal; Intraocular lens; Preloaded; Aphakic; Asqelio; aspicio; AST Products; ICARES
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- aspicio Monofocal IOL: A bi-aspheric monofocal IOL is implanted through preloaded IOL Delivery System in the capsular bag in the posterior chamber of the eye during cataract surgery
  Interventions: Device: aspicio Monofocal IOL

INTERVENTIONS:
Device: aspicio Monofocal IOL — A bi-aspheric monofocal IOL is implanted through preloaded IOL Delivery System in the capsular bag in the posterior chamber of the eye during cataract surgery
  Other Names: aspicio Monofocal; Asqelio Monofocal; ASPP60Y; ASP60Y; QPIO103Y; QLIO103Y

SUMMARY:
This is an observational, single-center, non-control, open-label post-marketing study. Patients implanted with an aspicio™ Monofocal Intraocular Lens will be scheduled for a follow-up visit at least 3 months after the surgery to undergo a routine basic ophthalmological examination.

DETAILED DESCRIPTION:
This is an observational, single-center, non-control, open-label post-marketing study. Patients implanted with an aspicio™ Monofocal Intraocular Lens will be scheduled for a single visit in the facilities of Chang Gung University Hospital at least 3 months after the surgery. Patients will undergo a routine basic ophthalmological examination.

Additionally, and retrospectively, the patients' medical records will be reviewed to obtain information on visual acuity and adverse events at postoperative visit carried out 1 month after surgery.

The data corresponding to the preoperative values of corneal curvature (flat meridian, curved meridian and axes), axial length measured by biometry, visual acuity and those corresponding to the implanted IOL will also be collected from the medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older who have been implanted with aspicio™ monofocal intraocular lens in at least 1 eye
2. Willingness to cooperate with and complete all post-operative visits
3. Ability to comprehend and sign an informed consent

Exclusion Criteria:

1. Any pathology that could reduce Visual Acuity (VA) (including amblyopia, severe corneal dystrophy, diabetic retinopathy, extremely narrow anterior chamber depth, microphthalmos, clinically significant macular/RPE changes, retinal detachment, corneal transplant, chronic sever uveitis, choroidal hemorrhage, recurrent severe inflammation of the anterior or posterior segment of unknown etiology, iris neovascularization, medically controlled or uncontrolled glaucoma, clinically significant macular degeneration, or diagnosis of pseudoexfoliation).
2. Previous ocular surgery (including YAG-laser) or trauma
3. Clinically significant irregular astigmatism
4. Concomitant severe eye disease
5. Pregnant or lactating
6. Any other ocular or systemic condition which, in the opinion of the investigator, should exclude the subject from the study
7. Concurrent participation in another drug or device investigation
8. May be expected to require other ocular surgery during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female adult patients who have been implanted with aspicio™ monofocal intraocular lens in at least 1 eye
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CDVA | 3 months after implantation
  Photopic monocular best corrected distance visual acuity (CDVA), 400cm
Defocus curve | 3 months after implantation
  Photopic monocular defocus curve, -4.0 D ~ +2.0 D

SECONDARY OUTCOMES:
UDVA | 3 months after implantation
  Photopic monocular uncorrected distance visual acuity (UDVA), 400cm
UIVA | 3 months after implantation
  Photopic monocular uncorrected intermediate visual acuity (UIVA), 60cm
CIVA | 3 months after implantation
  Photopic monocular corrected intermediate visual acuity (CIVA), 60cm
IOL glistening | 3 months after implantation
  IOL glistening observation
PCO | 3 months after implantation
  Posterior Capsular Opacification observation
Satisfaction questionnaire | 3 months after implantation
  Satisfaction questionnaire
AE | 3 months after implantation
  Signs of inflammation and AEs

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Shiou Hwang, MD, Principal Investigator — Chang Gung University Hospital
Locations (1):
- Chang Gung University Hospital, Taoyuan District, Guishan District, Taiwan

IPD SHARING:
Plan to Share IPD: No